CLINICAL TRIAL: NCT04457349
Title: Does Therapeutic Plasma Exchange Have A Role in Resistant Cytokine Storm State Of COVID-19 Infection?
Brief Title: Therapeutic Plasma Exchange in Resistant Cytokine Storm of COVID 19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, lecturer, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: plasma exchange in COVID 19
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Plasma Exchange; Plasmapheresis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic Plasma Exchange (TPE) (Experimental): Each patient will undergo two sessions. TPE will be done through filtration technique using a plasma filter at a dose of (1-1.5) plasma volume/session. Fresh frozen plasma or albumin 5% will be used to replace plasma.
  Interventions: Procedure: Therapeutic Plasma Exchange (TPE)

INTERVENTIONS:
Procedure: Therapeutic Plasma Exchange (TPE) — Treatment with Therapeutic Plasma Exchange (TPE)
  Other Names: plasmapheresis

SUMMARY:
This research is planned to illustrate the efficacy of Therapeutic Plasma Exchange (TPE) treatment in COVID-19 patients with resistant cytokine storm state.

DETAILED DESCRIPTION:
In early December 2019, several pneumonia cases of unknown origin were observed in Wuhan (China). A novel enveloped RNA β coronavirus was isolated and named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The new virus rapidly spread across China and worldwide. On March 11th 2020, the World Health Organization (WHO) declared coronavirus disease 2019 (COVID-19) a pandemic. As of 19June 2020, COVID-19 has been confirmed in 8,385,440 individuals globally with deaths reaching 450,686 with a morality of 5.37%. Egypt has 50,437 confirmed cases and 1938 deaths.

The virus mainly spreads through respiratory droplets from infected patients.The clinical spectrum of COVID-19 infection ranges from asymptomatic forms to severe pneumonia requiring hospitalization and isolation in critical care units with the need of mechanical ventilation due to acute respiratory distress syndrome (ARDS). Main symptoms include fever, fatigue and dry cough. Common laboratory findings include lymphopenia and elevated lactate dehydrogenase levels. Platelet count is usually normal or mildly decreased. C reactive protein (CRP) and erythrocyte sedimentation rate are usually increased while procalcitonin levels are normal and elevation of procalcitonin usually indicates secondary bacterial infection. Ferritin, D-dimer, and creatine kinase elevation is associated with severe disease. Chest computed tomographic scans show a typical pattern of bilateral patchy shadows or ground glass opacity.

Severe COVID-19 conditions are usually due to an aggressive inflammatory response known as "cytokine storm" that is characterized by the release of a large amount of pro-inflammatory cytokines. Lung injury, multiorgan failure, and unfavorable prognosis of severe COVID-19 infection have been attributed mainly to the cytokine storm state.

Many proinflammatory cytokines elevate in COVID-19 patients including IL-1, IL-6, IL-8, IL-10, tumour necrosis factor α (TNF-α) and interferon Ȣ(IFN-Ȣ) stimulating immune cells to invade sites of infection causing endothelial dysfunction, vascular damage, alveolar damage and ARDS. Cytokine storm has been reported in several viral infections including influenza H5N1 virus, influenza H1N1 virus, and the two coronaviruses highly related to COVID-19; "SARS-CoV" and "MERS-CoV".

Therapeutic approaches to manage the COVID-19 cytokine storm might provide an avenue to decrease the COVID-19 associated morbidity and mortality. Options include immunomodulators, cytokine antagonists and cytokine removal. Tocilizumab (IL-6 antagonist), Anakinra (antagonist of IL-1 β), TNF blockers, ruxolitinib (JAK1/2 inhibitor ), corticosteroids, intravenous immunoglobulins and therapeutic plasma exchange (TPE) have been used with variable efficacy.

Therapeutic plasma exchange can remove inflammatory factors, block the "cytokine storm", to reduce the damage of inflammatory response to the body. This therapy can be used for severe and critical patients in the early and middle stages of the disease. Patel and colleagues utilized TPE during the 2009 H1N1 influenza A outbreak in three pediatric patients presenting in a similar fashion to those seen with fulminant COVID-19 today. All three had full recovery from their illness after receiving rescue TPE. Adeli at al. used TPE as a rescue therapy in patients with severe forms of COVID-19 ( septic shock, ARDS ) with very good results. Out of 8 patients, 7 patients improved and one patient died. Zhang et al. also tried TPE in three COVID-19 patients who despite receiving antiviral treatment developed respiratory distress and levels of IL-6 increased rapidly. All patients improved clinically and radiologically with negative nucleic acid testing and were discharged 10-14 days later.

In Egypt, the first line drug to treat cytokine storm of COVID-19 is tocilizumab with good results. But a considerable percentage of patients do not respond to it leaving physicians with very limited options and usually patients deteriorated rapidly with high mortality. Based on the encouraging results of TPE in severe COVID-19 infections and the familiarity of the procedure, TPE could be a good option in those patients who do not respond to tocilizumab.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive patients (confirmed by PCR) with cytokine storm state who will not improve after two doses of tocilizumab.

  * Criteria of failure (resistance) to tocilizumab:

    1. Persistent high IL-6 and CRP.
    2. Persistent worsening of respiratory symptoms ( dyspnea, tachypnea, increased oxygen (O2) requirements or even need for mechanical ventilation).
    3. Partial arterial pressure of oxygen to fractional inspired concentration of oxygen (PaO2/FiO2) ratio < 150.
    4. Persistent fever (˃38.5°C) despite normal procalcitonin level.

Exclusion Criteria:

* Refractory septic shock:

( It is defined according to surviving sepsis campaign as the presence of hypotension with end organ dysfunction requiring high dose vasopressor support often greater than 0.5 µg/kg/min norepinephrine or equivalent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
mortality | 28 day
  Number of patients deaths of the total of patients included

SECONDARY OUTCOMES:
the mean time with oxygen therapy | through study completion, and average of 1 month
  to calculate the mean time with oxygen therapy
the mean time with Non-invasive mechanical ventilation | through study completion, and average of 1 month
  to calculate the mean time with Non-invasive mechanical ventilation
the mean time of intubation | through study completion, and average of 1 month
  to calculate the mean time of intubation
respiratory function parameters | through study completion, and average of 1 month
  To calculate the mean of PaO2/FiO2
respiratory function parameters | through study completion, and average of 1 month
  To calculate the mean of levels of oxygen saturation
radiological lung extension | through study completion, and average of 1 month
  to evaluate the lung extension of pneumonia
mean duration of hospitalization and ICU use | through study completion, and average of 1 month
  Days of hospitalization in survivors and/or days at ICU throughout the study
the requirement of additional organ support | through study completion, and average of 1 month
  Percentage of patients with dialysis
the levels of IL-6 | through study completion, and average of 1 month
  To evaluate the effect of TPE on the serum levels of inflammatory markers
Incidence of adverse events | through study completion, and average of 1 month
  To calculate the number of adverse events in patients with COVID-19 treated with TPE
time to reverse-transcriptase polymerase chain reaction (RT-PCR) virus negativity | through study completion, and average of 1 month
  To evaluate the time to RT-PCR virus negativity
the levels of CRP | through study completion, and average of 1 month
  To evaluate the effect of TPE on the serum levels of inflammatory markers
the levels of procalcitonin (PCT) | through study completion, and average of 1 month
  To evaluate the effect of TPE on the serum levels of inflammatory markers
levels of D-dimer | through study completion, and average of 1 month
  To evaluate the effect of TPE on the serum levels of inflammatory markers
levels of ferritin | through study completion, and average of 1 month
  To evaluate the effect of TPE on the serum levels of inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — Lecturer of Nephrology & Internal Medicine, Faculty of Medicine, Alexandria university, Egypt; montasser M zeid, MD, Study Chair — Professor of Nephrology & Internal Medicine, Faculty of Medicine, Alexandria university, Egypt; Akram M Fayed, MD, Study Chair — Professor of Critical Care Medicine, Faculty of Medicine, Alexandria university, Egypt; Ehab M El Reweny, MD, Study Chair — Assistant Professor of Critical Care Medicine, Faculty of Medicine, Alexandria university, Egypt; Nermine H Zakaria, MD, Study Chair — Professor of Clinical and Chemical Pathology Medicine, Faculty of Medicine, Alexandria university, Egypt; Ayman I Baess, MD, Study Chair — Assistant Professor of Chest Diseases, Faculty of Medicine, Alexandria university, Egypt
Locations (1):
- Faculty of Medicine, Alexandria university, Egypt, Alexandria, Egypt

REFERENCES:
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Singhal T. A Review of Coronavirus Disease-2019 (COVID-19). Indian J Pediatr. 2020 Apr;87(4):281-286. doi: 10.1007/s12098-020-03263-6. Epub 2020 Mar 13. PMID 32166607
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835
- [Background] Sun D, Li H, Lu XX, Xiao H, Ren J, Zhang FR, Liu ZS. Clinical features of severe pediatric patients with coronavirus disease 2019 in Wuhan: a single center's observational study. World J Pediatr. 2020 Jun;16(3):251-259. doi: 10.1007/s12519-020-00354-4. Epub 2020 Mar 19. PMID 32193831
- [Background] Kalaiyarasu S, Kumar M, Senthil Kumar D, Bhatia S, Dash SK, Bhat S, Khetan RK, Nagarajan S. Highly pathogenic avian influenza H5N1 virus induces cytokine dysregulation with suppressed maturation of chicken monocyte-derived dendritic cells. Microbiol Immunol. 2016 Oct;60(10):687-693. doi: 10.1111/1348-0421.12443. PMID 27730669
- [Background] Channappanavar R, Perlman S. Pathogenic human coronavirus infections: causes and consequences of cytokine storm and immunopathology. Semin Immunopathol. 2017 Jul;39(5):529-539. doi: 10.1007/s00281-017-0629-x. Epub 2017 May 2. PMID 28466096
- [Background] Ye Q, Wang B, Mao J. The pathogenesis and treatment of the ;Cytokine Storm' in COVID-19. J Infect. 2020 Jun;80(6):607-613. doi: 10.1016/j.jinf.2020.03.037. Epub 2020 Apr 10. PMID 32283152
- [Background] Patel P, Nandwani V, Vanchiere J, Conrad SA, Scott LK. Use of therapeutic plasma exchange as a rescue therapy in 2009 pH1N1 influenza A--an associated respiratory failure and hemodynamic shock. Pediatr Crit Care Med. 2011 Mar;12(2):e87-9. doi: 10.1097/PCC.0b013e3181e2a569. PMID 20453703
- [Background] Adeli SH, Asghari A, Tabarraii R, Shajari R, Afshari S, Kalhor N, Vafaeimanesh J. Therapeutic plasma exchange as a rescue therapy in patients with coronavirus disease 2019: a case series. Pol Arch Intern Med. 2020 May 29;130(5):455-458. doi: 10.20452/pamw.15340. Epub 2020 May 7. No abstract available. PMID 32380821
- [Background] Zhang L, Zhai H, Ma S, Chen J, Gao Y. Efficacy of therapeutic plasma exchange in severe COVID-19 patients. Br J Haematol. 2020 Aug;190(4):e181-e183. doi: 10.1111/bjh.16890. Epub 2020 Jun 12. No abstract available. PMID 32453903
- [Background] Bassi E, Park M, Azevedo LC. Therapeutic strategies for high-dose vasopressor-dependent shock. Crit Care Res Pract. 2013;2013:654708. doi: 10.1155/2013/654708. Epub 2013 Sep 15. PMID 24151551